CLINICAL TRIAL: NCT02283047
Title: Effects on Blood Pressure, Cardiorespiratory Condition and Cardiovascular Risk of Different Aerobic Exercise Programs With Nutritional Interventions in Hypertensive and Overweight People.
Brief Title: Effects of Different Aerobic Exercise Programs With Nutritional Interventions in Hypertensive and Overweight People
Acronym: EXERDIET-HTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of the Basque Country (UPV/EHU) (Other)
Collaborators: IMQ-Igualatorio Médico Quirúrgico, Vitoria-Gasteiz (Araba/Álava) (Unknown); Servicios Tecnológicos de Tecnalia (Unknown); Hospital Comarcal Santiago Apostol, Miranda de Ebro (Burgos) (Unknown)
Responsible Party: Principal Investigator, SARA MALDONADO-MARTIN, Dr. Sara Maldonado-Martin PhD, University of the Basque Country (UPV/EHU)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHU14/08
Record Dates: First submitted 2014-10-21; First posted 2014-11-05 (Estimated); Last update posted 2017-06-23 (Actual); Status verified 2017-06

CONDITIONS: Hypertension; Overweight; Sedentary
Keywords: cardiovascular risk, obesity, interval training, diet
MeSH Terms: conditions — Hypertension; Overweight; Sedentary Behavior; Obesity | interventions — Diet; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CONTROL GROUP-DIET (Active Comparator): Hypocaloric diet intervention with no supervised exercise intervention
  Interventions: Behavioral: DIET
- DIET & MODERATE CONTINUOUS TRAINING (Experimental): Intervention with hypocaloric diet and supervised moderate continuous exercise training (60-80%HRpeak). High volume training (45 minutes in progression from 20 min)
  Interventions: Behavioral: DIET & MODERATE CONTINUOUS TRAINING
- DIET & HIGH VOLUME HIIT (Experimental): Intervention with hypocaloric diet and supervised high intensity interval training (85-95%HRpeak). High volume training (45 minutes in progression from 20 min)
  Interventions: Behavioral: DIET & HIGH VOLUME HIIT
- DIET & LOW VOLUME HIIT (Experimental): Intervention with hypocaloric diet and supervised high intensity interval training (85-95%HRpeak). Low volume training (20 min)
  Interventions: Behavioral: DIET & LOW VOLUME HIIT

INTERVENTIONS:
Behavioral: DIET — Lifestyle intervention through hypocaloric diet
  Other Names: CONTROL GROUP
  Arms: CONTROL GROUP-DIET
Behavioral: DIET & MODERATE CONTINUOUS TRAINING — Lifestyle intervention through hypocaloric diet and exercise at moderate intensity (60-80%peakHR) continuous mode, and high volume (45 min).
  Other Names: MCT
  Arms: DIET & MODERATE CONTINUOUS TRAINING
Behavioral: DIET & HIGH VOLUME HIIT — Lifestyle intervention through hypocaloric diet and exercise at high intensity (80-95%peakHR) interval mode, and high volume (45 min).
  Other Names: HV-HIIT
  Arms: DIET & HIGH VOLUME HIIT
Behavioral: DIET & LOW VOLUME HIIT — Lifestyle intervention through diet and exercise at high intensity (80-95%peakHR) interval mode, and low volume (20 min).
  Other Names: LV-HIIT
  Arms: DIET & LOW VOLUME HIIT

SUMMARY:
Obesity and arterial hypertension (HTN) frequently coexist in the same patient. Moreover, the concept that obesity and HTN can be additive in terms of cardiovascular rist is widely accepted. Yet, clinical decision-making in obese patients is complicated by a surprising lack of evidence on the relative importance of obesity and HTN treatment and its efficacy and safety. Lifestyle interventions are the mainstay of obesity management programs and are also advocated in the prevention and treatment of HTN. Physical exercise and diet are recommended to prevent and control obesity and HTN. Aerobic exercise is firmly established as an effective measure for lowering blood pressure and reducing cardiovascular risk. However, there is no agreement about the optimal dose of frequency, intensity, duration and type of exercise. Therefore, the aims of the study are: 1) to assess the changes in selected parameters of blood pressure, cardiorespiratory fitness, body composition and biological markers brought about by a period of 16-week of different aerobic exercise programs with hypocaloric diet for overweight or obesity and primary hypertensive adults, and 2) to examine the effect of six months detraining subsequent to intervention. Secondary objectives are to examine the additional effect of the intervention on physical activity behavior and health-related quality of life.

DETAILED DESCRIPTION:
METHODOLOGY: participants will perform a ramp incremental cardiopulmonary exercise bike test before, after 16-week of follow-up, and after 6-month detraining period (with no intervention only recommendations). After inclusion criteria they will be randomized to four parallel groups: 1) control group with only hypocaloric diet intervention and lifestyle recommendations; 2) Moderate (HR values between VT1 and VT2 or 50-75% of HR reserve) continuous exercise and high volume (from 20 to 45min) group and hypocaloric diet intervention; 3) high intensity (HR values up to VT2 to peak intensity or ≥76% to <100 % of HR reserve) interval training and high-volume (from 20 to 45min) group alternating high and moderate intensities at different protocols and hypocaloric diet intervention; and 4) high-intensity interval training and low-volume (20min) group alternating high and moderate intensities at different protocolsand hypocaloric diet intervention.

ELIGIBILITY:
Inclusion Criteria:

* older than 18yr old and less than 70yr old
* overweight (BMI >25)
* primary hypertension
* low-moderate cardiovascular risk
* not diet treatment
* sedentary behavior
* availability to exercise two days a week.

Exclusion Criteria:

* secondary hypertension
* pulmonary disorder
* neurological deficit
* physical incapacity to exercise
* to exercise frequently
* pregnancy or breastfeeding
* left ventricular hypertrophy
* more than three cardiovascular risk factors

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Actual)
Dates: Start 2015-01; Primary Completion 2016-06 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Blood pressure | 16-weeks
  Ambulatory Blood Pressure Monitoring- 24 hours-Systolic and diastolic blood pressure

SECONDARY OUTCOMES:
Health related Quality of life (QoL) | 16-weeks
  Questionnaire SF-36
Incremental shuttle walk test (ISWT) | 16-weeks
  Field test
Ventilatory threshold (VT) | 16-weeks
  the VT is the 'point of transition between predominantly aerobic energy production to anaerobic energy production
Biochemical variables | 16-weeks
  Glucose, Insulin, Leptin, Adiponectin,Total-Cholesterol, HDL-cholesterol, LDL-cholesterol, Triglycerides, C-reactive protein, aspartate transaminase, alanine transaminase, gamma-glutaryl transferase, Fibrinogen Uric acid
Physical activity and sedentary behavior | 16-weeks
  Accelerometry and The International Physical Activity Questionnaires
Peak Oxygen Uptake (VO2peak) | 16-weeks
  Cardiovascular peak aerobic capacity
Anthropometry | 16-weeks
  Body mass, body mass index, waist-hip ratio

CONTACTS AND LOCATIONS:
Overall Officials: SARA MALDONADO-MARTIN, PhD, Principal Investigator — University of the Basque Country (UPV/EHU)
Locations (1):
- Faculty of Physical Activity and Sport Sciences, Vitoria-Gasteiz, Araba/alava, Spain

REFERENCES:
- [Background] Mancia G, De Backer G, Dominiczak A, Cifkova R, Fagard R, Germano G, Grassi G, Heagerty AM, Kjeldsen SE, Laurent S, Narkiewicz K, Ruilope L, Rynkiewicz A, Schmieder RE, Boudier HA, Zanchetti A; ESH-ESC Task Force on the Management of Arterial Hypertension. 2007 ESH-ESC Practice Guidelines for the Management of Arterial Hypertension: ESH-ESC Task Force on the Management of Arterial Hypertension. J Hypertens. 2007 Sep;25(9):1751-62. doi: 10.1097/HJH.0b013e3282f0580f. No abstract available. PMID 17762635
- [Background] Agueda M, Lasa A, Simon E, Ares R, Larrarte E, Labayen I. Association of circulating visfatin concentrations with insulin resistance and low-grade inflammation after dietary energy restriction in Spanish obese non-diabetic women: role of body composition changes. Nutr Metab Cardiovasc Dis. 2012 Mar;22(3):208-14. doi: 10.1016/j.numecd.2010.06.010. Epub 2010 Oct 14. PMID 20951014
- [Background] Cornelissen VA, Goetschalckx K, Verheyden B, Aubert AE, Arnout J, Persu A, Rademakers F, Fagard RH. Effect of endurance training on blood pressure regulation, biomarkers and the heart in subjects at a higher age. Scand J Med Sci Sports. 2011 Aug;21(4):526-34. doi: 10.1111/j.1600-0838.2010.01094.x. Epub 2010 Mar 10. PMID 20459467
- [Background] Gibala MJ, Little JP, Macdonald MJ, Hawley JA. Physiological adaptations to low-volume, high-intensity interval training in health and disease. J Physiol. 2012 Mar 1;590(5):1077-84. doi: 10.1113/jphysiol.2011.224725. Epub 2012 Jan 30. PMID 22289907
- [Background] Jimenez-Pavon D, Ortega FB, Artero EG, Labayen I, Vicente-Rodriguez G, Huybrechts I, Moreno LA, Manios Y, Beghin L, Polito A, De Henauw S, Sjostrom M, Castillo MJ, Gonzalez-Gross M, Ruiz JR; HELENA Study Group. Physical activity, fitness, and serum leptin concentrations in adolescents. J Pediatr. 2012 Apr;160(4):598-603.e2. doi: 10.1016/j.jpeds.2011.09.058. Epub 2011 Nov 13. PMID 22082954
- [Background] Molmen-Hansen HE, Stolen T, Tjonna AE, Aamot IL, Ekeberg IS, Tyldum GA, Wisloff U, Ingul CB, Stoylen A. Aerobic interval training reduces blood pressure and improves myocardial function in hypertensive patients. Eur J Prev Cardiol. 2012 Apr;19(2):151-60. doi: 10.1177/1741826711400512. Epub 2011 Mar 4. PMID 21450580
- [Derived] Gorostegi-Anduaga I, Tous-Espelosin M, Maldonado-Martin S. Does greater adherence to a healthy dietary pattern correspond to a better body composition and cardiorespiratory fitness in adults with overweight and primary hypertension? Data from the EXERDIET-HTA study. Blood Press Monit. 2025 Jun 1;30(3):104-108. doi: 10.1097/MBP.0000000000000731. PMID 39436237
- [Derived] Gorostegi-Anduaga I, Corres P, MartinezAguirre-Betolaza A, Perez-Asenjo J, Aispuru GR, Fryer SM, Maldonado-Martin S. Effects of different aerobic exercise programmes with nutritional intervention in sedentary adults with overweight/obesity and hypertension: EXERDIET-HTA study. Eur J Prev Cardiol. 2018 Mar;25(4):343-353. doi: 10.1177/2047487317749956. Epub 2018 Jan 9. PMID 29313359
- See also: Given the ever increasing prevalence of hypertension in the United States and the issues involved in treating cases of resistant and complex hypertension, the Leadership of the American Society of Hypertension, Inc. (ASH) recognizes that hypertension can — http://www.ash-us.org/